CLINICAL TRIAL: NCT03981055
Title: Parkinson's Disease: Enhancing Physical Therapy With Brain Stimulation for Treating Postural Instability.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director, Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital & Massachusetts General Hospital, Harvard Medical School, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018P002733; R44NS110237 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-06-10 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS and Active TUS (Experimental): Active tDCS and Active TUS for 20 min
  Interventions: Device: Active Comparator: Active tDCS and Active TUS; Other: Physical Therapy
- Sham TDCS and Sham TUS (Sham Comparator): Sham TDCS and Sham TUS for 20 min
  Interventions: Device: Sham Comparator: Sham TDCS and Sham TUS; Other: Physical Therapy

INTERVENTIONS:
Device: Active Comparator: Active tDCS and Active TUS — Device: Transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Arms: Active tDCS and Active TUS
Device: Sham Comparator: Sham TDCS and Sham TUS — Device: SHAM Comparator Device: transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Arms: Sham TDCS and Sham TUS
Other: Physical Therapy — All subjects will enroll in a conventional PT balance and gait focused training program, and will receive PT 3x/week over the two weeks of stimulation for 45 minutes following the stimulation sessions when applicable. (And during the biweekly sessions for Phase II)

SUMMARY:
This trial aims to understand the mechanism and to test whether transcranial direct current stimulation (tDCS) combined with transcranial ultrasound (TUS) (tDCS+TUS) combined with physical therapy (PT) will induce significant therapeutic effects in postural instability in Parkinson's disease (PT) patients. The investigators designed a double-blinded, placebo controlled, randomized study to investigate the effects of 2 weeks of TDCS+TUS on postural instability in PD patients receiving PT. (Followed by biweekly sessions for 2 more weeks in Phase II)

DETAILED DESCRIPTION:
Current treatments for Parkinson's Disease (PD), including pharmacological (levodopa) and surgical (DBS) methods, have limited impact on postural instability. Physical therapy (PT) for PD is becoming increasingly used as a means to induce benefits on patient balance. However, limits in efficacy and consistency still exist. In this study, the investigators will test the effects of TDCS+TUS combined with PT on postural instability of PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of "probable" or "possible" PD, as defined by the current clinical criteria (Gelb D, Oliver E, Gilman S. Diagnostic Criteria for Parkinson's Disease. Arch Neurol.1999;56:33-39) as confirmed by co-investigator neurologist, or confirmation via medical records or a letter from patient physician;
2. Complaints about balance impairment or postural instability due to PD (self-report);
3. Age from 40 to 90 years old;
4. Taking stable medications for PD for at least 30 days.

Exclusion Criteria:

1. Features suggestive of other causes of parkinsonism/Parkinson's-plus syndromes;
2. History of deep brain stimulation or brain ablation surgeries, malignant mass brain lesions;
3. History of schizophrenia, bipolar illness; history of alcohol/drug abuse within the past 6 months;
4. Need for rapid clinical response due to conditions such as initiation, psychosis, or suicidality;
5. Contraindications to transcranial brain stimulation or TUS, i.e. metal in the head, implanted brain medical devices, etc.;
6. Unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, uncompensated pulmonary disease, or chronic obstructive pulmonary disease);
7. Pregnancy.
8. Epilepsy or disorders that significantly increase likelihood of seizures including: severe traumatic brain injury, congenital birth defects leading to seizures, brain tumor, metabolic disorders associated with seizures, intracranial or subarachnoid hemorrhage, and nonlacunar strokes.
9. Recent (<= 2 months) or planned enrollment in an additional physician prescribed physical therapy program during their time in the trial.
10. Presence of another disorder that might have a significant impact on balance (as assessed by a co-investigator neurologist).
11. Bed or wheelchair-bound

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS and Active TUS: Active tDCS and Active TUS for 20 min
  Active Comparator: Active tDCS and Active TUS: Device: Transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Physical Therapy: All subjects will enroll in a conventional PT balance and gait focused training program, and will receive PT 3x/week over the two weeks of stimulation for 45 minutes following the stimulation sessions when applicable. (And during the biweekly sessions for Phase II)
- Sham TDCS and Sham TUS: Sham TDCS and Sham TUS for 20 min
  Sham Comparator: Sham TDCS and Sham TUS: Device: SHAM Comparator Device: transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Physical Therapy: All subjects will enroll in a conventional PT balance and gait focused training program, and will receive PT 3x/week over the two weeks of stimulation for 45 minutes following the stimulation sessions when applicable. (And during the biweekly sessions for Phase II)
Period: Overall Study
Arm/Group | Active tDCS and Active TUS | Sham TDCS and Sham TUS
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline for randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS and Active TUS | Sham TDCS and Sham TUS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.35 (9.33) | 68.2 (9.13) | 66.77 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 13 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Unified Parkinson's Disease Rating Scale (UPDRS) Part III
Description: Motor function was assessed using the Unified Parkinson's Disease Rating Scale (UPDRS) Part III - Motor Examination, which measures tremor, rigidity, bradykinesia, postural instability, and gait.
  Scores range from 0 to 108, where higher scores indicate worse motor impairment (i.e., lower scores represent better motor function).
Time Frame: Change from baseline to Day 14 (end of stimulation treatment).
Population: Intention-to-treat population: all randomized participants with Parkinson's disease
Measure: Mean (Standard Error); unit: Scores on a scale (UPDRS).
Arm/Group | Active tDCS and Active TUS | Sham TDCS and Sham TUS
Number analyzed (Participants) | 20 | 20
Scores on a scale (UPDRS). | 4.42 (0.42) | 0.12 (0.43)

ADVERSE EVENTS:
Time Frame: 14 weeks.
Description: Adverse effects were collected with a questionnaire for adverse effects.
Arm/Group | Active tDCS and Active TUS | Sham TDCS and Sham TUS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS and Active TUS (N=20) | Sham TDCS and Sham TUS (N=20)
Tingling (Skin and subcutaneous tissue disorders) | 20 (181) | 13 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03981055/Prot_SAP_002.pdf